CLINICAL TRIAL: NCT05027425
Title: Durvalumab (MEDI4736) and Tremelimumab for Hepatocellular Carcinoma in Patients Listed for a Liver Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Davendra Sohal (Other)
Responsible Party: Sponsor-Investigator, Davendra Sohal, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-GI-21-01
Record Dates: First submitted 2021-08-17; First posted 2021-08-30 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma; Cirrhosis; Portal Hypertension
Keywords: Transplant
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Hypertension, Portal | interventions — durvalumab; tremelimumab; Liver Transplantation

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label, Phase II, multicenter clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Durvalumab + Tremelimumab + Liver Transplant (Experimental): Patients will be treated with the immunotherapy combination for up to 4 months. After a minimum 28 day washout, they will undergo locoregional therapy per institutional standards. Eventually, after a minimum 72-day washout from the end of immunotherapy, they will undergo liver transplant.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Procedure: Liver Transplant

INTERVENTIONS:
Drug: Durvalumab — 1500 mg IV, Q4W
  Other Names: MEDI4736
Drug: Tremelimumab — 300 mg IV, 1 dose on day 1 of only the first cycle
Procedure: Liver Transplant — minimum 72-day washout from the end of immunotherapy, patients will undergo liver transplant.

SUMMARY:
Immunotherapy can safely downstage patients and achieve durable systemic disease control to improve clinical outcomes in HCC patients undergoing liver transplant.

DETAILED DESCRIPTION:
ESR-20-21010 is a single-arm, open-label, Phase II, multicenter clinical trial designed to evaluate the safety and efficacy of durvalumab and tremelimumab for the treatment of hepatocellular carcinoma (HCC) patients who have cirrhosis or portal hypertension and are evaluated by institutional Liver Transplant team and deemed eligible for transplant.

The key eligibility requirements include HCC, Child-Pugh score of up to 7, and ECOG PS of 0 or 1.

Patients will be treated with the immunotherapy combination for up to 4 months. After a minimum 28 day washout, they will undergo locoregional therapy per institutional standards. Eventually, after a minimum 72-day washout from the end of immunotherapy, they will undergo liver transplant.

The primary endpoint is proportion of patients experiencing post-transplant rejection (within 30 days of transplant). A total of 30 patients are to be enrolled, to allow at least 20 transplants for adequate primary endpoint analysis. An interim analysis after 10 patients will be performed to ensure safety. If there are untoward safety signals, study modification/discontinuation will be discussed.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular carcinoma, diagnosed either by biopsy or by combination of cirrhosis and imaging criteria (contrast-enhanced CT or MRI).
2. Tumor confined to liver with no vascular invasion and no evidence of extrahepatic disease.
3. Patient evaluated by institutional Liver Transplant team and listed for transplant.
4. At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion (TL) at baseline. Tumor assessment by computed tomography (CT) scan or magnetic resonance imaging (MRI) must be performed within 28 days prior to randomization.
5. No prior therapy for HCC at any time.
6. Age ≥18 years at the time of study entry.
7. ECOG score of 0 or 1
8. Child-Pugh Score of 5, 6, or 7
9. Body weight >30 kg
10. Patients must have adequate organ and marrow function as defined in protocol
11. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Extrahepatic disease.
2. Variceal bleeding during 3 months prior to registration.
3. Any autoimmune disease deemed a risk in the setting of immunotherapy per treating physician's judgment.
4. Any other illness or patient condition deemed a medical or logistical barrier for protocol therapy per treating physician's judgment.
5. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
6. Participation in another clinical study with an investigational product during the last 12 months Patients who have received other investigational agents previously who are no longer receiving these investigational agents may be eligible at the discretion of the PI.
7. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
8. History of allogenic organ transplantation.
9. History of another primary malignancy except for:

   1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   3. Adequately treated carcinoma in situ without evidence of disease
10. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
12. History of leptomeningeal carcinomatosis
13. History of active primary immunodeficiency
14. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
15. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
16. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine while receiving IP and up to 30 days after the last dose of IP.
17. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab + tremelimumab combination therapy.
18. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
19. Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
20. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2030-12-07 (Estimated)

PRIMARY OUTCOMES:
Cellular rejection rates | Up to 30 days post transplant
  To assess the safety of immunotherapy for treatment of HCC in patients listed for a liver transplant, with respect to cellular rejection rates

SECONDARY OUTCOMES:
Adverse events during treatment, and graft loss and mortality rates | Treatment, and up to 30 days post transplant
  To assess the safety of immunotherapy for treatment of HCC in patients listed for a liver transplant, with respect to adverse events during treatment, and graft loss and mortality rates up to 30 days after transplant;
Radiologic responses via RECIST 1.1 and/or mRECIST | Survival follow up will continue for 5 years after end of Treatment
  To assess the efficacy of immunotherapy for treatment of HCC in patients listed for a liver transplant, with respect to radiologic responses
Pathologic responses via explanted liver assessment | Survival follow up will continue for 5 years after end of Treatment
  To assess the efficacy of immunotherapy for treatment of HCC in patients listed for a liver transplant, with respect to Pathologic responses
Recurrence-free survival and overall survival outcomes based on survival follow up reporting | Survival follow up will continue for 5 years after end of Treatment
  To assess the efficacy of immunotherapy for treatment of HCC in patients listed for a liver transplant, with respect to Survival outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Davendra Sohal, MD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - Simmons Comprehensive Cancer Center UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided